CLINICAL TRIAL: NCT00381940
Title: A Phase II Study of Bortezomib (Velcade, PS-341) in Combination With Ifosfamide/Vinorelbine in Pediatric Patients and Young Adults With Refractory/Recurrent Hodgkin Disease
Brief Title: Bortezomib, Ifosfamide, and Vinorelbine Tartrate in Treating Young Patients With Hodgkin's Lymphoma That is Recurrent or Did Not Respond to Previous Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01063; NCI-2009-01063 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000500142; AHOD0521 (Other: Children's Oncology Group); AHOD0521 (Other: CTEP); U10CA098543 (NIH); NCT01648439 (obsolete NCT alias)
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Results first posted 2014-04-10 (Estimated); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Adult Lymphocyte Depletion Hodgkin Lymphoma; Adult Lymphocyte Predominant Hodgkin Lymphoma; Adult Mixed Cellularity Hodgkin Lymphoma; Adult Nodular Lymphocyte Predominant Hodgkin Lymphoma; Adult Nodular Sclerosis Hodgkin Lymphoma; Childhood Lymphocyte Depletion Hodgkin Lymphoma; Childhood Lymphocyte Predominant Hodgkin Lymphoma; Childhood Mixed Cellularity Hodgkin Lymphoma; Childhood Nodular Lymphocyte Predominant Hodgkin Lymphoma; Childhood Nodular Sclerosis Hodgkin Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent/Refractory Childhood Hodgkin Lymphoma; Stage I Adult Hodgkin Lymphoma; Stage I Childhood Hodgkin Lymphoma; Stage II Adult Hodgkin Lymphoma; Stage II Childhood Hodgkin Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Childhood Hodgkin Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Childhood Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Recurrence | interventions — Ifosfamide; indolepropanol phosphate; Bortezomib; Vinorelbine; Filgrastim; Granulocyte Colony-Stimulating Factor

ARMS (1):
- Treatment (enzyme inhibitor therapy, chemotherapy) (Experimental): Patients receive ifosfamide IV continuously over days 1-4, vinorelbine ditartrate IV over 6-10 minutes on days 1 and 5, bortezomib IV on days 1, 4, and 8, and filgrastim (G-CSF) IV or subcutaneously beginning on day 6 and continuing until blood counts recover or PBSC are harvested. Treatment repeats every 21 days for up to 2 or 4 courses in the absence of disease progression or unacceptable toxicity.
  Patients undergo autologous PBSC harvesting according to institutional guidelines after the second course of therapy.
  Interventions: Drug: ifosfamide; Drug: bortezomib; Drug: vinorelbine tartrate; Biological: filgrastim

INTERVENTIONS:
Drug: ifosfamide — Given IV
  Other Names: Cyfos; Holoxan; IFF; IFX; IPP
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Drug: vinorelbine tartrate — Given IV
  Other Names: Eunades; navelbine ditartrate; NVB; VNB
Biological: filgrastim — Given IV or SC
  Other Names: G-CSF; Neupogen

SUMMARY:
This phase II trial studies the side effects and efficacy of bortezomib with ifosfamide and vinorelbine in children and young adults with Hodgkin's lymphoma that was recurrent or did not respond to previous therapy. Bortezomib is an inhibitor of protein degradation. Bortezomib degrades short-lived regulatory proteins in the cell, and has been reported to increase the tumor cells. Bortezomib may increase the effectiveness of ifosfamide and vinorelbine (two standard drugs given to children with Hodgkin Lymphoma that has come back after initial treatment) by making cancer cells more sensitive to effectiveness of standard chemotherapy by preventing anti-death responses in these drugs. Giving bortezomib together with ifosfamide and vinorelbine tartrate should kill more cancer cells than are killed with ifosfamide and vinorelbine alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the efficacy and safety of bortezomib (as a chemosensitizing agent) in pediatric patients and young adults with primary refractory Hodgkin's lymphoma (HL) or HL in first relapse.

II. Determine the response rate in patients treated with bortezomib, ifosfamide, and vinorelbine ditartrate (vinorelbine tartrate) (IVB) and compare the response rate to the historical response rate in patients treated with ifosfamide and vinorelbine ditartrate alone.

SECONDARY OBJECTIVES:

I. Determine the overall response rate (complete and partial response) and induction success rate after 2 or 4 courses of therapy and the reinduction rate (complete response) after 4 courses of therapy.

II. Determine the proportion of patients able to mobilize sufficient hematopoietic stem cells (CD34+) after 2 courses of IVB.

OUTLINE: This is a multicenter, open-label, pilot study.

Patients receive ifosfamide intravenously (IV) continuously over days 1-4, vinorelbine tartrate IV over 6-10 minutes on days 1 and 5, and bortezomib intravenously on days 1, 4, and 8, and filgrastim (G-CSF) by vein or subcutaneously beginning on day 6 and continuing until blood counts recover or peripheral blood stem cells (PBSC) are harvested. Treatment cycles repeat every 21 days for up to 2 or 4 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo autologous PBSC harvesting according to institutional guidelines after the second course of therapy.

After completion of study treatment, patients are followed every 6 months for 2 years and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Hodgkin's lymphoma at time of relapse or disease progression, meeting all of the following criteria:

  * Stage I-IV disease
  * No morphologically unclassifiable disease
* Meets 1 of the following criteria:

  * Mixed cellularity
  * Lymphocytic depletion (LD)
  * LD, diffuse fibrosis
  * LD, reticular
  * Lymphocyte predominance (LP)
  * LP, diffuse
  * LP, nodular
  * Nodular sclerosis (NS)
  * NS, cellular phase
  * NS, lymphocytic predominance
  * NS, mixed cellularity
  * NS, LD
  * Not otherwise specified
* Primary refractory disease OR disease in first relapse, except for the following:

  * Patients who achieved a complete response after treatment on protocol COG-AHOD0431 who experience a biopsy-proven recurrence after doxorubicin hydrochloride, vincristine, prednisone, and cyclophosphamide without involved-field radiotherapy
  * Patients on the observation-only arm of protocol COG-AHOD0431
* Any measurable, focal mass lesion of a visceral organ (e.g., liver, spleen, or kidney)
* Patients with metastatic disease to bone marrow and granulocytopenia, anemia, and/or thrombocytopenia are allowed provided both of the following criteria are met:

  * Platelet count ≥ 20,000/mm³ (platelet transfusion allowed)
  * Hemoglobin ≥ 8 g/dL (packed red blood cell transfusion allowed)
* Karnofsky performance status (PS) 60-100% (for patients > 16 years of age) OR Lanksy PS 60-100% (for patients =< 16 years of age)
* Life expectancy >= 2 months
* Absolute neutrophil count >= 1,000/mm^3
* Platelet count >= 75,000/mm^3 (transfusion independent) (for patients with no bone marrow involvement)
* Creatinine =< 1.5 times upper limit of normal (ULN)
* Creatinine clearance or radioisotope glomerular filtration rate >= 70 mL/min/1.73 m^2
* AST and ALT =< 2.5 times ULN
* Bilirubin =< 1.5 times ULN
* Shortening fraction >= 27% by echocardiogram OR LVEF >= 50% by gated radionuclide study
* Patients with a seizure disorder are eligible if on a nonenzyme-inducing anticonvulsant and seizures are well controlled
* No CNS toxicity > grade 2
* No serious intercurrent illnesses
* No known hypersensitivity to E. coli-derived proteins, filgrastim (G-CSF), or any component of the study drugs
* No peripheral neuropathy > grade 1
* No known hypersensitivity to bortezomib, boron, or mannitol
* No other concurrent chemotherapy or immunomodulating agents (including steroids)

  * Concurrent corticosteroids allowed for treatment or prophylaxis of anaphylactic reactions
  * No dexamethasone or aprepitant as an antiemetic
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Recovered from prior therapy
* No prior bortezomib or other proteasome inhibitors
* At least 3 weeks since prior chemotherapy (4 weeks for nitrosoureas)
* More than 14 days since prior investigational drugs
* No concurrent enzyme inducing anticonvulsants that alter p450 metabolism, including phenytoin, carbamazepine, phenobarbital, or other anticonvulsants

  * Benzodiazepine or gabapentin allowed

Max Age: 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2007-01; Primary Completion 2008-06 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terzah Horton, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Horton TM, Drachtman RA, Chen L, Cole PD, McCarten K, Voss S, Guillerman RP, Buxton A, Howard SC, Hogan SM, Sheehan AM, Lopez-Terrada D, Mrazek MD, Agrawal N, Wu MF, Liu H, De Alarcon PA, Trippet TM, Schwartz CL. A phase 2 study of bortezomib in combination with ifosfamide/vinorelbine in paediatric patients and young adults with refractory/recurrent Hodgkin lymphoma: a Children's Oncology Group study. Br J Haematol. 2015 Jul;170(1):118-22. doi: 10.1111/bjh.13388. Epub 2015 Apr 1. PMID 25833390

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Ifosfamide, Vinorelbine, Bortezomib): This was a single arm study that treated all patients with ifosfamide, vinorelbine, and bortezomib. Patients received ifosfamide IV (3000 mg/m2/day) continuously over days 1-4, vinorelbine ditartrate IV (25 mg/m2/dose) over 6-10 minutes on days 1 and 5, bortezomib IV (1.2 mg/m2/dose) on days 1, 4, and 8, and filgrastim (G-CSF) IV or subcutaneously beginning on day 6 and continuing until blood counts recover or PBSC are harvested. Treatment cycle repeats every 21 days for up to 2 or 4 courses in the absence of disease progression or unacceptable toxicity.
  Patients undergo autologous PBSC harvesting according to institutional guidelines after the second course of therapy.
  ifosfamide: Given IV
  bortezomib: Given IV
  vinorelbine ditartrate: Given IV
  filgrastim: Given IV or SC
Period: Overall Study
Arm/Group | Treatment (Ifosfamide, Vinorelbine, Bortezomib)
Started | 26
Completed | 21
Not Completed | 5
Not completed — Lack of Efficacy | 3
Not completed — Protocol Violation | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ifosfamide, Vinorelbine, Bortezomib)
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.9 (2.6)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 18
  More than one race | 0
  Unknown or Not Reported | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23
  Australia | 1
  Canada | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR)
Description: CR is defined as at least 80% reduction in the sum of the products of the perpendicular diameters of each of the nodal masses or return to normal size, along with negative nuclear medicine imaging.
Time Frame: After 2 cycles of treatment
Population: Analysis population includes all patients evaluable for tumor response. Three enrolled patients are excluded: 1 ineligible, 1 who was removed from treatment after 1 dose of bortezomib, and 1 who received only 1/3 dose of bortezomib in cycle 1 and part of cycle 2 due to pharmacy error.
Measure: Number; unit: participants
Arm/Group | Treatment (Ifosfamide, Vinorelbine, Bortezomib)
Number analyzed (Participants) | 23
participants
  With CR | 2
  Without CR | 21

2. Secondary Outcome: Number of Participants With Grade 3 or 4 Toxicity
Description: Grade 3 and 4 non-hematologic toxicity during protocol therapy. The number of patients that experience CTC Version 4 grade 3 or higher non-hematologic at any time during protocol therapy
Time Frame: 4 weeks following completion of therapy
Population: 25 patients reported, 1 ineligible patient not included in adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ifosfamide, Vinorelbine, Bortezomib)
Number analyzed (Participants) | 25
Participants | 9

3. Secondary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: After 2 cycles and 4 cycles
Population: There were 23 patients evaluable after 2 cycles and 12 patients evaluable after 4 cycles. 1 patient was excluded after cycle 2 and cycle 4 due to pharmacy error. 2 patients were excluded after cycle 2 due to ineligibility and removal from treatment after 1 dose of bortezomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ifosfamide, Vinorelbine, Bortezomib)
Number analyzed (Participants) | 23
Participants
  Overall Response Rate (After 2 cycles) | 19
  Overall Response Rate (After 4 cycles): number analyzed (Participants) | 12
  Overall Response Rate (After 4 cycles) | 12

4. Secondary Outcome: Induction Success Rate
Description: Induction success is defined as achieving CR or PR without a targeted primary toxicity. Primary toxicity includes toxic death (which is any death predominantly attributable to treatment-related toxicities or complications, occurring during or within one month of the completion of therapy), Non-hematologic grades 3 or 4 toxicities attributable to drug (with the specific exclusion of 1) Grade 3 or 4 nausea or vomiting, 2) grade 3 transaminases (AST/ALT) elevations which return to < grade 1 prior to the time of the next treatment course, 3) grade 3 or 4 fever or infection, and 4) Grade 3 mucositis.) and Hematologic toxicity (Delay of >2 weeks in the start of re-induction cycle 2 or in hematologic recovery after cycle 2 secondary to severe myelosuppression, infection, or sepsis.)
Time Frame: After 2 cycles and 4 cycles
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ifosfamide, Vinorelbine, Bortezomib)
Number analyzed (Participants) | 23
Participants
  Induction Success Rate (After 2 cycles) | 19
  Induction Success Rate (After 4 cycles): number analyzed (Participants) | 12
  Induction Success Rate (After 4 cycles) | 12

5. Secondary Outcome: Rate of Successful PBSC Harvest
Description: Success is defined as the ability to harvest 2x10^6 CD34+ cells/kg within 5 collection days.
Time Frame: After 2 cycles
Population: Analysis population includes all patients evaluable after cycle 2. Six enrolled patients are excluded: 1 ineligible, 1 who was removed from treatment after 1 dose of bortezomib, and 1 who received only 1/3 dose of bortezomib in cycle 1 and part of cycle 2 due to pharmacy error, 3 who did not have recorded data
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ifosfamide, Vinorelbine, Bortezomib)
Number analyzed (Participants) | 20
Participants | 19

6. Secondary Outcome: Biological Markers
Description: Assessing baseline NF-kB protein levels in tumor tissue
Time Frame: Before, during, and after treatment
Population: Corresponding data were not collected
Arm/Group | Treatment (Ifosfamide, Vinorelbine, Bortezomib)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: 25 patients reported, 1 ineligible patient not included in adverse events.
Arm/Group | Treatment (Ifosfamide, Vinorelbine, Bortezomib)
Serious Adverse Events (participants affected / at risk) | 4/25
Other Adverse Events (participants affected / at risk) | 18/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ifosfamide, Vinorelbine, Bortezomib) (N=25)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ifosfamide, Vinorelbine, Bortezomib) (N=25)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Death NOS (General disorders) | 3 (3)
Catheter related infection (Infections and infestations) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 7 (7)
Urinary tract infection (Infections and infestations) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (4)
Neutrophil count decreased (Investigations) | 6 (6)
Platelet count decreased (Investigations) | 3 (3)
White blood cell decreased (Investigations) | 5 (5)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neuralgia (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less